CLINICAL TRIAL: NCT02927275
Title: Cognition in Motion: Attitudes, Utilization, and Cognitive Impact of Low Intensity Exercise Among Medical Students
Brief Title: Cognition in Motion
Acronym: CIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Cecilia Valdes, MD, Associate Professor-Obstetrics & Gynecology, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H-31608
Record Dates: First submitted 2016-10-01; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Cognitive Performance During Physical Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standing Modality (Experimental): Performance on computerized cognitive tests while standing at a desk. Experimental: Standing Modality
  Interventions: Behavioral: Experimental: Standing Modality
- Biking Modality (Experimental): Performance on computerized cognitive tests while biking at user's preferred speed on stationary bicycle. Experimental: Biking Modality
  Interventions: Behavioral: Experimental: Biking Modality
- Walking Modality (Experimental): Performance on computerized cognitive tests while walking at 1mph. Experimental: Walking Modality
  Interventions: Behavioral: Experimental: Walking Modality
- Seated Modality (Other): Performance on computerized cognitive tests while sitting. No Intervention: Seated Modality
  Interventions: Behavioral: No Intervention: Seated Modality

INTERVENTIONS:
Behavioral: Experimental: Standing Modality — Cognitive performance when standing
  Arms: Standing Modality
Behavioral: Experimental: Biking Modality — Cognitive performance when biking slowly
  Arms: Biking Modality
Behavioral: Experimental: Walking Modality — Cognitive performance when walking at 1mph
  Arms: Walking Modality
Behavioral: No Intervention: Seated Modality — Cognitive performance when sitting.
  Arms: Seated Modality

SUMMARY:
The purpose of this study is to evaluate the effect of low-intensity exercise on cognitive functioning during activity. Evaluation was accomplished by having participants perform standardized cognitive tests while in three forms of low-intensity exercise and then comparing results to performance when sitting.

DETAILED DESCRIPTION:
While studies have demonstrated the beneficial effects of exercise, even when low-intensity, on physical health, investigations into cognitive performance during these periods of activity are increasing in number. For changes in the workplace to occur, data needs to show that mental processing is not compromised while engaging in low-intensity exercise.

In this current study, participants, after giving written consent, performed quantitative, computer-based cognitive tests to evaluate for differences in performance between active and sedentary conditions. The participants engaged in four activity modalities: sitting, standing, biking slowly on a stationary bicycle, and walking at 1mph. The validated tests used were immediate and delayed verbal recall, the color-word test based on the Stroop test, and the "n-back" test. Responses were scored according to both the speed in answering along with accuracy on each test. From the scores generated, effect sizes were calculated for sitting and compared to effect sizes for cumulative activity stations for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Student at Baylor College of Medicine
* Able to perform low-intensity exercise

Exclusion Criteria:

* Not a student at Baylor College of Medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cognitive Testing Performance | Starting in April 2012, participant enrollment was open for 41 months with data collection occurring immediately at the time of testing with no need for follow-up outcome measurements.
  Scores generated from cognitive testing

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia T Valdes, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine-Department of Obstetrics & Gynecology, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual performance on testing rounds was incorporated into cumulative statistical analysis and will not be made public.

REFERENCES:
- [Background] Ogden CL, Carroll MD, Fryar CD, Flegal KM. Prevalence of Obesity Among Adults and Youth: United States, 2011-2014. NCHS Data Brief. 2015 Nov;(219):1-8. PMID 26633046
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of regular physical activity among adults--United States, 2001 and 2005. MMWR Morb Mortal Wkly Rep. 2007 Nov 23;56(46):1209-12. PMID 18030281
- [Background] U.S. Department of Health and Human Services. 2008 physical activity guidelines for Americans. 2008; http://health.gov/PAGuidelines/pdf/paguide.pdf. Accessed May 22, 2016.
- [Background] Haskell WL. Physical activity by self-report: a brief history and future issues. J Phys Act Health. 2012 Jan;9 Suppl 1:S5-10. doi: 10.1123/jpah.9.s1.s5. PMID 22287448
- [Background] Bey L, Hamilton MT. Suppression of skeletal muscle lipoprotein lipase activity during physical inactivity: a molecular reason to maintain daily low-intensity activity. J Physiol. 2003 Sep 1;551(Pt 2):673-82. doi: 10.1113/jphysiol.2003.045591. Epub 2003 Jun 18. PMID 12815182
- [Background] van der Berg JD, Stehouwer CD, Bosma H, van der Velde JH, Willems PJ, Savelberg HH, Schram MT, Sep SJ, van der Kallen CJ, Henry RM, Dagnelie PC, Schaper NC, Koster A. Associations of total amount and patterns of sedentary behaviour with type 2 diabetes and the metabolic syndrome: The Maastricht Study. Diabetologia. 2016 Apr;59(4):709-18. doi: 10.1007/s00125-015-3861-8. Epub 2016 Feb 2. PMID 26831300
- [Background] Dunstan DW, Salmon J, Owen N, Armstrong T, Zimmet PZ, Welborn TA, Cameron AJ, Dwyer T, Jolley D, Shaw JE; AusDiab Steering Committee. Associations of TV viewing and physical activity with the metabolic syndrome in Australian adults. Diabetologia. 2005 Nov;48(11):2254-61. doi: 10.1007/s00125-005-1963-4. Epub 2005 Oct 7. PMID 16211373
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825
- [Background] Wennberg P, Boraxbekk CJ, Wheeler M, Howard B, Dempsey PC, Lambert G, Eikelis N, Larsen R, Sethi P, Occleston J, Hernestal-Boman J, Ellis KA, Owen N, Dunstan DW. Acute effects of breaking up prolonged sitting on fatigue and cognition: a pilot study. BMJ Open. 2016 Feb 26;6(2):e009630. doi: 10.1136/bmjopen-2015-009630. PMID 26920441
- [Background] Reiff C, Marlatt K, Dengel DR. Difference in caloric expenditure in sitting versus standing desks. J Phys Act Health. 2012 Sep;9(7):1009-11. doi: 10.1123/jpah.9.7.1009. PMID 22971879
- [Background] Cox RH, Guth J, Siekemeyer L, Kellems B, Brehm SB, Ohlinger CM. Metabolic cost and speech quality while using an active workstation. J Phys Act Health. 2011 Mar;8(3):332-9. doi: 10.1123/jpah.8.3.332. PMID 21487132
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- [Background] LeBlanc AG, Spence JC, Carson V, Connor Gorber S, Dillman C, Janssen I, Kho ME, Stearns JA, Timmons BW, Tremblay MS. Systematic review of sedentary behaviour and health indicators in the early years (aged 0-4 years). Appl Physiol Nutr Metab. 2012 Aug;37(4):753-72. doi: 10.1139/h2012-063. PMID 22765839
- [Background] Buckley JP, Hedge A, Yates T, Copeland RJ, Loosemore M, Hamer M, Bradley G, Dunstan DW. The sedentary office: an expert statement on the growing case for change towards better health and productivity. Br J Sports Med. 2015 Nov;49(21):1357-62. doi: 10.1136/bjsports-2015-094618. Epub 2015 Jun 1. PMID 26034192
- [Background] Francois ME, Baldi JC, Manning PJ, Lucas SJ, Hawley JA, Williams MJ, Cotter JD. 'Exercise snacks' before meals: a novel strategy to improve glycaemic control in individuals with insulin resistance. Diabetologia. 2014 Jul;57(7):1437-45. doi: 10.1007/s00125-014-3244-6. Epub 2014 May 10. PMID 24817675
- [Background] Baldo JV, Delis D, Kramer J, Shimamura AP. Memory performance on the California Verbal Learning Test-II: findings from patients with focal frontal lesions. J Int Neuropsychol Soc. 2002 May;8(4):539-46. doi: 10.1017/s135561770281428x. PMID 12030307
- [Background] Stroop J. Studies of interference in serial verbal reactions. Journal of Experimental Psychology. 1935;18:643-62.
- [Background] KIRCHNER WK. Age differences in short-term retention of rapidly changing information. J Exp Psychol. 1958 Apr;55(4):352-8. doi: 10.1037/h0043688. No abstract available. PMID 13539317
- [Background] Donner Y. Computational Approaches to Scaling Up Experimental Science. Stanford University Libraries: Computer Science, Stanford University; 2015.
- [Background] Ebara T, Kubo T, Inoue T, Murasaki GI, Takeyama H, Sato T, Suzumura H, Niwa S, Takanishi T, Tachi N, Itani T. Effects of adjustable sit-stand VDT workstations on workers' musculoskeletal discomfort, alertness and performance. Ind Health. 2008 Oct;46(5):497-505. doi: 10.2486/indhealth.46.497. PMID 18840942
- [Background] Dutta N, Koepp GA, Stovitz SD, Levine JA, Pereira MA. Using sit-stand workstations to decrease sedentary time in office workers: a randomized crossover trial. Int J Environ Res Public Health. 2014 Jun 25;11(7):6653-65. doi: 10.3390/ijerph110706653. PMID 24968210
- [Background] Thorp AA, Kingwell BA, Owen N, Dunstan DW. Breaking up workplace sitting time with intermittent standing bouts improves fatigue and musculoskeletal discomfort in overweight/obese office workers. Occup Environ Med. 2014 Nov;71(11):765-71. doi: 10.1136/oemed-2014-102348. Epub 2014 Aug 28. PMID 25168375
- [Background] Labonte-LeMoyne E. Santhanam R., Leger P.M., Courtemanche F., Fredette M., Senecal S. The delayed effect of treadmill desk usage on recall and attention. Computers in Human Behavior. 2015;46:1-5.
- [Background] Commissaris DA, Konemann R, Hiemstra-van Mastrigt S, Burford EM, Botter J, Douwes M, Ellegast RP. Effects of a standing and three dynamic workstations on computer task performance and cognitive function tests. Appl Ergon. 2014 Nov;45(6):1570-8. doi: 10.1016/j.apergo.2014.05.003. Epub 2014 Jun 17. PMID 24951234
- [Background] Thompson WG, Levine JA. Productivity of transcriptionists using a treadmill desk. Work. 2011;40(4):473-7. doi: 10.3233/WOR-2011-1258. PMID 22130064
- [Background] Bantoft C, Summers MJ, Tranent PJ, Palmer MA, Cooley PD, Pedersen SJ. Effect of Standing or Walking at a Workstation on Cognitive Function: A Randomized Counterbalanced Trial. Hum Factors. 2016 Feb;58(1):140-9. doi: 10.1177/0018720815605446. Epub 2015 Sep 24. PMID 26408647
- [Background] John D, Bassett D, Thompson D, Fairbrother J, Baldwin D. Effect of using a treadmill workstation on performance of simulated office work tasks. J Phys Act Health. 2009 Sep;6(5):617-24. doi: 10.1123/jpah.6.5.617. PMID 19953838
- [Background] Ohlinger CM, Horn TS, Berg WP, Cox RH. The effect of active workstation use on measures of cognition, attention, and motor skill. J Phys Act Health. 2011 Jan;8(1):119-25. doi: 10.1123/jpah.8.1.119. PMID 21297192
- [Background] Alderman BL, Olson RL, Mattina DM. Cognitive function during low-intensity walking: a test of the treadmill workstation. J Phys Act Health. 2014 May;11(4):752-8. doi: 10.1123/jpah.2012-0097. PMID 25078520
- [Background] Swagerman SC, de Geus EJ, Koenis MM, Hulshoff Pol HE, Boomsma DI, Kan KJ. Domain dependent associations between cognitive functioning and regular voluntary exercise behavior. Brain Cogn. 2015 Jul;97:32-9. doi: 10.1016/j.bandc.2015.04.001. Epub 2015 May 24. PMID 25956142
- [Background] Tudor-Locke C, Schuna JM Jr, Frensham LJ, Proenca M. Changing the way we work: elevating energy expenditure with workstation alternatives. Int J Obes (Lond). 2014 Jun;38(6):755-65. doi: 10.1038/ijo.2013.223. Epub 2013 Nov 28. PMID 24285335
- [Background] Pontifex MB, Hillman CH. Neuroelectric and behavioral indices of interference control during acute cycling. Clin Neurophysiol. 2007 Mar;118(3):570-80. doi: 10.1016/j.clinph.2006.09.029. Epub 2006 Nov 13. PMID 17095295
- [Background] Davranche K, Hall B, McMorris T. Effect of acute exercise on cognitive control required during an Eriksen flanker task. J Sport Exerc Psychol. 2009 Oct;31(5):628-39. doi: 10.1123/jsep.31.5.628. PMID 20016112
- [Background] Straker L, Levine J, Campbell A. The effects of walking and cycling computer workstations on keyboard and mouse performance. Hum Factors. 2009 Dec;51(6):831-44. doi: 10.1177/0018720810362079. PMID 20415158
- [Background] Larson MJ, LeCheminant JD, Hill K, Carbine K, Masterson T, Christenson E. Cognitive and typing outcomes measured simultaneously with slow treadmill walking or sitting: implications for treadmill desks. PLoS One. 2015 Apr 15;10(4):e0121309. doi: 10.1371/journal.pone.0121309. eCollection 2015. PMID 25874910
- [Background] Levine JA, Miller JM. The energy expenditure of using a "walk-and-work" desk for office workers with obesity. Br J Sports Med. 2007 Sep;41(9):558-61. doi: 10.1136/bjsm.2006.032755. Epub 2007 May 15. PMID 17504789
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] MacEwen BT, MacDonald DJ, Burr JF. A systematic review of standing and treadmill desks in the workplace. Prev Med. 2015 Jan;70:50-8. doi: 10.1016/j.ypmed.2014.11.011. Epub 2014 Nov 28. PMID 25448843